CLINICAL TRIAL: NCT00161928
Title: A Randomized, Open-Label Trial of NeisVac-C Vaccine to Evaluate Immunological Interference With Hepatitis B, Inactivated Polio and Acellular Pertussis Vaccines in Healthy Infants
Brief Title: Study of NeisVac-C Vaccine to Evaluate Immunological Interference With Hepatitis B, Inactivated Polio and Acellular Pertussis Vaccines in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 216
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Meningitis, Meningococcal
Keywords: Meningococcal Vaccine; Meningococcal Meningitis, Serogroup C; Neisseria Meningitidis
MeSH Terms: conditions — Meningitis, Meningococcal

INTERVENTIONS:
Biological: Group C Meningococcal Polysaccharide-Tetanus Toxoid Conjugate Vaccine (GCMP-TT)

SUMMARY:
The primary aim of the study is to show that NeisVac-C does not influence the seroconversion rates induced by hepatitis B (Hep B), inactivated polio (IPV) and acellular pertussis (aP) vaccines in infants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers infants, aged 2 to 6 months
* Clinically healthy, (i.e. the physician would have no reservations vaccinating with a meningococcal C vaccine outside the scope of a clinical trial)
* Parent(s)/legal guardian understands the study and has provided written informed consent for his/her infant's study participation
* Parent(s)/legal guardian and infant will be available for the duration of the study

Exclusion Criteria:

* History of any vaccine-related contraindicating event (e.g. anaphylaxis)
* Rash or other dermatological condition at the injection site which could interfere with injection site reaction monitoring or lead to a dermatological reaction
* Subjects who have received or will receive other vaccine(s) ± 30 days before or after the study period
* Concurrent participation in or previous participation in a clinical trial with an investigational medicinal product
* Subjects who suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids, chemotherapeutics) that can be expected to influence immunological functions
* Subjects who have previously received a vaccination against Hep B or meningococcal C
* Subjects who have received banked human blood or immunoglobulins within one month of study entry

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330
Dates: Start 2002-04; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (14):
- Austria (2):
  - Freistädter Strasse 290, Linz
  - Grieskirchner Strasse 17, Wels
- Germany (12):
  - Neuschwansteinstrasse 5, Augsburg
  - Marktplatz 3, Bad Saulgau
  - Hasenheide 66, Berlin
  - Hauptstrasse 9, Bietigheim-Bissingen
  - Rheinstrasse13, Ettenheim
  - Solothurner Strasse 2, Heilbronn
  - Haupstrasse 240, Kehl
  - Löpsinger Strasse 8, Nördlingen
  - Tuchbergstrasse 2, Oberndorf / Neckar
  - Asternweg 11a, Offenburg
  - Falkensteiner Strasse 24, Roding
  - Broner Platz 6, Weingarten